CLINICAL TRIAL: NCT04351958
Title: An Augmented Reality Videogame for Alcohol Use Prevention and Harm
Brief Title: An Augmented Reality Videogame for Alcohol Use Prevention and Harm Reduction in Teens
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000027338; No NIH funding (Other: 11.09.23)
Record Dates: First submitted 2020-02-20; First posted 2020-04-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Prevention; Harm Reduction
Keywords: videogame; augmented reality
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Intervention Model Description: Pre-Post Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented Reality ("No Time Wasted") (Experimental)
  Interventions: Behavioral: Experimental: Augmented Reality ("No Time Wasted")

INTERVENTIONS:
Behavioral: Experimental: Augmented Reality ("No Time Wasted") — "No Time Wasted" will be an innovative, immersive intervention using novel technology that will captivate the target audience with narrative and gaming elements to scaffold the educational message.

SUMMARY:
The goal of this research study is to develop the AR-based alcohol use prevention and harm reduction intervention, "No Time Wasted", with the further aim of conducting a pre-post pilot study to assess whether the game reduce risk behaviors associated with alcohol use, whilst also increasing knowledge about some of the following topics: BAC, standard drink sizes, signs of alcohol poisoning. The intervention will also seek to encourage bystander intervention to assist fictional characters in need of help due to overdrinking.

DETAILED DESCRIPTION:
Specific Aim #1: DEVELOPMENT: A prototype of an augmented reality (AR) videogame intervention for alcohol use prevention and harm reduction in adolescents aged 16-18. Input from 4 focus groups of 5 adolescents each (n = 20), and the extant literature will inform the development of the AR videogame intervention, "No Time Wasted".

Specific Aim #2: PILOT EVALUATION: Conduct a pre-post pilot study with 20 teens ages 16-18 collecting assessment data at baseline and immediately following gameplay to assess

"No Time Wasted" will be an innovative, immersive intervention using novel technology that will captivate the target audience with narrative and gaming elements to scaffold the educational message. The proposed research will be conducted in two phases. Phase I consists of: (a) the development of the prototype using input from 4 focus groups of 5 adolescents each (n = 20), aged 16-18 and the extant literature (Specific Aim #1). In Phase II will consisted of a pre-post pilot study with 20 teens ages 16-18 collecting assessment data at baseline and immediately following gameplay to assess 1) the intervention's acceptability and feasibility by collecting quantitative and qualitative data on teens' satisfaction and gameplay experience of the intervention, and 2) the preliminary impact of the intervention on knowledge, intentions, perceptions, attitudes, social norms, self-efficacy and behaviors related to alcohol use and harm reduction.

Conduct focus groups to gather data to develop the AR videogame prototype, "No Time Wasted": Four focus groups will be conducted (5 adolescents each) to collect feedback on the game content, narrative, characters, and gameplay mechanics. To facilitate the discussions, visual tools (e.g., storyboards, pictures) will be used. The focus groups will be conducted according to standard dual-facilitator procedures. The four focus groups will be adequate to achieve thematic saturation. The focus groups will be conducted such that ideas and themes from one discussion inform discussion topics and prompts used in the next focus group. Audio recordings of each session will be transcribed, reviewed, and discussed by the research team to refine the videogame intervention. As a part of the game development and with parental permission, selected students will be invited to the Yale recording studio on campus to provide voices for the videogame characters.

Conduct a pre-post pilot study: This study will enroll 20 adolescents ages 16-18 using a pre/post design to evaluate the feasibility, acceptability, and preliminary efficacy of the AR videogame prototype. Participants will accumulate between 1- 1.5 hours of game play over 2 sessions (approximately one week, meeting twice). This total duration and number of sessions is consistent with those found in effective alcohol harm reduction and prevention interventions, which range from 10 minutes to 4 hours, and with the amount of time adolescents play videogames. Participants will have a 15-10 min break in the middle of each session and will be instructed that they may take additional breaks as needed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 16-18 years of age and currently enrolled in high school
* Speak English
* Able to play an AR videogame (willing use an AR headset for 30-45 minutes/session to play the game for the pilot study).
* Eligibility will be determined by the research team.

Exclusion Criteria:

-

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To determine participants' satisfaction and gameplay experience | End of gameplay - 2 hours
  Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 5 items on game experience and satisfaction from items designed for a previous videogame study on sexual risk reduction in young adolescents (e.g., "I would tell my friends to play this game," Questions have 5-point Likert-type choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 response choices ranging from very unlikely to very likely.

SECONDARY OUTCOMES:
Behaviors with alcohol pretest | Baseline
  To determine the baseline alcohol use behavior and attitudes--pretest survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then play the videogame intervention. The 5 questions from the 2019 Youth Risk Behavior Survey (YRBS) that pertain to alcohol consumption will be used to assess participant alcohol use behavior. These items relate to frequency of drinking in the past 30 days (0-30), frequency of binge drinking in the past 30 days (0-20), and the maximum number of drinks consumed in a row in the last 30 days (1-10).
Knowledge of alcohol pre-test | Baseline
  To determine the impact of an AR harm reduction and prevention videogame prototype, FREEZE!, on participants' knowledge about alcohol - Pre-test survey.
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), before playing the videogame intervention. A 12-item true/false/not sure block of questions will be developed to assess knowledge about alcohol information such as symptoms of alcohol poisoning, standard drink sizes, social host laws, common alcohol and drug interactions, and myths and misconceptions about alcohol.
Knowledge of alcohol post-test | End of gameplay - 2 hours
  To determine the impact of an AR harm reduction and prevention videogame prototype, FREEZE!, on participants' knowledge about alcohol - Post-test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after playing the videogame intervention. A 12-item true/false/not sure block of questions will be developed to assess knowledge about alcohol information such as symptoms of alcohol poisoning, standard drink sizes, social host laws, common alcohol and drug interactions, and myths and misconceptions about alcohol.
Intentions, attitudes, and social norms pre-test | Baseline
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), before playing the videogame intervention.The Brief Adolescent Alcohol Expectancy Questionnaire (AEQ-AB) is designed to measure the degree to which individuals expect alcohol to produce a variety of general and specific effects. Research with the AEQ indicates a consistent relationship between alcohol expediencies and alcohol consumption, alcohol abuse and behavior while drinking. This questionnaire has 7 items that address intentions about drinking, attitudes towards both positive and negative components of alcohol consumption, and questions that address peer alcohol expectations and related social norms.
Intentions, attitudes, and social norms post-test | End of gameplay - 2 hours
  Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after playing the videogame intervention.The Brief Adolescent Alcohol Expectancy Questionnaire (AEQ-AB) is designed to measure the degree to which individuals expect alcohol to produce a variety of general and specific effects. Research with the AEQ indicates a consistent relationship between alcohol expediencies and alcohol consumption, alcohol abuse and behavior while drinking. This questionnaire has 7 items that address intentions about drinking, attitudes towards both positive and negative components of alcohol consumption, and questions that address peer alcohol expectations and related social norms.
Self-efficacy to refuse pre-test | Baseline
  Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software), before playing the videogame intervention.The 9-item Drinking Refusal Self-Efficacy Question are Shortened Revised Adolescent version (DRSEQ-SRA) is a shortened version of the DRSEQ-RA. It measures levels of drinking refusal self-efficacy, or confidence in an adolescent's ability to resist alcohol in cued situations. Responses are rated on a 6-point Likert scale (1 = I am very sure I could NOT resist drinking to 6 = I am very sure I could resist drinking). It comprises three subscales: Emotional relief refusal self-efficacy (3 items, e.g., 'When I feel sad'); Opportunistic refusal self-efficacy (3 items, e.g., 'When I am listening to music or reading'); Social pressure refusal self-efficacy (3 items, e.g., 'When my friends are drinking').
Self-efficacy to refuse post-test | End of gameplay - 2 hours
  Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after playing the videogame intervention.The 9-item Drinking Refusal Self-Efficacy Question are Shortened Revised Adolescent version (DRSEQ-SRA) is a shortened version of the DRSEQ-RA. It measures levels of drinking refusal self-efficacy, or confidence in an adolescent's ability to resist alcohol in cued situations. Responses are rated on a 6-point Likert scale (1 = I am very sure I could NOT resist drinking to 6 = I am very sure I could resist drinking). It comprises three subscales: Emotional relief refusal self-efficacy (3 items, e.g., 'When I feel sad'); Opportunistic refusal self-efficacy (3 items, e.g., 'When I am listening to music or reading'); Social pressure refusal self-efficacy (3 items, e.g., 'When my friends are drinking').

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hieftje, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided